CLINICAL TRIAL: NCT06170268
Title: Alzheimer's National Registry for Treatment and Diagnostics
Brief Title: Alzheimer's National Registry for Treatment and Diagnostics(ALZ-NET)
Acronym: ALZ-NET
Status: Recruiting | Type: Observational
Sponsor: Alzheimer's Disease and Related Disorders Association, Inc (Other)
Collaborators: American College of Radiology (Other); The Critical Path Institute (Unknown); Brown University (Other); American Society of Neuroradiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALZ-NET
Record Dates: First submitted 2022-07-07; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Trials; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Biospecimen collection and retention will be included in a future protocol amendment. Detail will be provided once available and approved by the IRB of record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Not Applicable/Open Label Registry: ALZ-NET is a growing network of sites that follow participants over time with an expandable platform, allowing for the collection of real-world data from enrolled patients being evaluated for or receiving any novel FDA-approved Alzheimer's disease therapies. ALZ-NET is treatment agnostic. Drug treatment dosage, frequency and duration will be guided by FDA label and clinician judgment as part of treatment and patient management.
  Interventions: Other: Routine Care Documentation

INTERVENTIONS:
Other: Routine Care Documentation — Routine Care Documentation

SUMMARY:
The Alzheimer's Network for Treatment and Diagnostics (ALZ-NET) will collect longitudinal clinical and safety data for enrolled patients being evaluated for or treated with novel FDA-approved Alzheimer's disease (AD) therapies. ALZ-NET is a longitudinal registry with an expandable platform, designed to grow with scientific and medical advancements. As new treatments are approved and implemented in care, ALZ-NET will track the long-term health outcomes associated with their use in a real-world setting. ALZ-NET is a resource for evidence gathering, information sharing and education across clinical and research communities, encouraging innovative research and supporting opportunities to improve clinical care delivery. All participating physicians and site staff will complete comprehensive training to ensure adherence of data requirements and registry timelines.

DETAILED DESCRIPTION:
ALZ-NET is collecting longitudinal clinical and safety data for enrolled patients that are being evaluated for or being treated with novel FDA-approved AD therapies. ALZ-NET is a longitudinal registry with an expandable platform, designed to grow with scientific and medical advancements. As new treatments are approved and implemented in care, ALZ-NET will track the long-term health outcomes associated with their use in a real-world setting. ALZ-NET aims to assess the clinical course of people from a variety of backgrounds and communities, to achieve representativeness beyond the populations historically enrolled in clinical trials. ALZ-NET will be a resource for evidence gathering, information sharing, and education across clinical and research communities, encouraging innovative, inclusive research and supporting opportunities to improve clinical care delivery.

ALZ-NET will align with the following objectives:

* Collect baseline and longitudinal patient data, including measures of cognition, function, and long-term safety.
* Collect and archive diagnostic, neuroimaging, genetic and fluid biomarkers.
* Track health outcomes and resource utilization through existing databases.
* Share deidentified data, images and biosamples with the research community and other stakeholders.

All participating physicians and site staff will complete comprehensive training to ensure adherence of data requirements and registry timelines. ALZ-NET will collect longitudinal data through site submitted case report forms and payer claims. Additional objectives of ALZ-NET are to establish a biorepository of plasma, CSF and DNA samples and to archive brain images from participants who consent to these optional elements.

In addition to the aims and objectives outlined within this protocol, ALZ-NET will serve as a backbone registry and platform for collection of regulatory grade data and collaboration with affiliated studies. Affiliated studies are thoroughly reviewed by the ALZ-NET Steering Committee before receiving affiliation approval. ALZ-NET will allow for seamless co enrollment of participants that are being evaluated for or receiving a novel FDA-approved treatment for AD. This collaboration structure is designed to reduce the operational burden of participating sites and patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient or patient's legally authorized representative (LAR) or proxy (e.g., spouse or legal guardian) has the ability to understand the purpose and risks of ALZ-NET and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local patient privacy regulations.
* Patient is at least 18 years of age at the time of informed consent.
* Patient has a diagnosis of MCI or dementia with clinical suspicion of AD as contributing pathology and (1) is being evaluated for treatment or, (2) will be initiating treatment, or (3) has already initiated treatment with novel FDA-approved AD therapies in real-world clinical practice.
* If treatment is initiated at the time of consent, patient meets appropriate label requirements and treatment follows appropriate use recommendations for novel FDA-approved AD therapy/therapies.
* Patient's treating clinician has made the decision to provide clinical care or treatment prior to patient consent and independently of the purpose of ALZ-NET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults of all racial and ethnic backrounds that have memory concerns and/ or may have diagnosis of Alzheimer's disease (AD) and has been identified by an approved site investigator (as defined by protocol) to be appropriate for treatment with novel FDA-approved therapies in real world clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether FDA-approved treatments improve health outcomes (as measured by slowing of cognitive decline) over time in a real-world population in broad clinical settings. | 2 years
  The primary measure of cognitive status will be the overall score of Montreal Cognitive Assessment (MoCA). MoCA is measured on a scale of 0 to 30 with higher scores indicating better cognitive function.
Evaluate whether FDA-approved treatments improve health outcomes (as measured by slowing of cognitive decline) over time in a real-world population in broad clinical settings. | 2 years
  The primary measures of cognitive status will be the overall score of the Mini Mental State Examination (MMSE). MMSE is measured on a scale of 0 to 30 with higher scores indicating better cognitive function.
Evaluate whether FDA-approved treatments improve health outcomes (as measured by slowing of functional decline) over time in a real-world population in broad clinical settings. | 2 years
  The primary measure of functional status will be the overall score of the Functional Activities Questionnaire (FAQ). FAQ is measured on a scale of 0 to 30 with higher scores indicating more impaired function.
Evaluate safety outcomes of FDA-approved treatments over time in a real-world population in broad clinical settings. | 2 years
  The measures of safety will be summaries of rates of adverse events over time. Specific safety outcomes of interest include amyloid related imaging abnormalities (ARIA)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Rabinovici, MD, Principal Investigator — University of California, San Francisco; Maria C Carillo, PhD, Principal Investigator — Alzheimer's Association; Michael S Rafii, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- Full List of Active Sites, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
ALZ-NET is committed to providing investigators in academia and industry an opportunity to access data collected as part of the network for purposes that are consistent with the goals of ALZ-NET. ALZ-NET archives the clinical and image data obtained as part of its research activity. This archive can be used for secondary research studies, to guide further drug or technology development, and for educational purposes. Access to CMS claims data used in ALZ-NET is handled separately and requires permission from CMS. Any individual or entity may submit a request for the clinical data, image data, or images linked to clinical data archived by ALZ-NET. The Network will provide requesters the raw data as it is archived in the database. However, requesters can specify subsets of data they desire using the annotated elements from the case report forms. The identity (and identifiable information) of network participants, sites and investigators will not be provided to requesters.
Access Criteria: The application forms for requesting archived clinical and image data is available on upon request. Requests for access to the ALZ-NET archive should be sent to alz-net@acr.org. Before indicating in a grant proposal that clinical and/or image data archived by ALZ-NET will be used to conduct the proposed research, an investigator should submit a request and obtain written approval from ALZ-NET prior to submitting the grant proposal. ALZNET treats such requests as it does any other.

REFERENCES:
- [Background] 2022 Alzheimer's disease facts and figures. Alzheimers Dement. 2022 Apr;18(4):700-789. doi: 10.1002/alz.12638. Epub 2022 Mar 14. PMID 35289055
- [Background] Rajan KB, Weuve J, Barnes LL, McAninch EA, Wilson RS, Evans DA. Population estimate of people with clinical Alzheimer's disease and mild cognitive impairment in the United States (2020-2060). Alzheimers Dement. 2021 Dec;17(12):1966-1975. doi: 10.1002/alz.12362. Epub 2021 May 27. PMID 34043283
- [Background] Guerreiro R, Bras J. The age factor in Alzheimer's disease. Genome Med. 2015 Oct 20;7:106. doi: 10.1186/s13073-015-0232-5. PMID 26482651
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] 2021 Alzheimer's disease facts and figures. Alzheimers Dement. 2021 Mar;17(3):327-406. doi: 10.1002/alz.12328. Epub 2021 Mar 23. PMID 33756057
- See also: ALZ-NET Website — https://www.alz.org/professionals/health-systems-clinicians/management/alzheimers-network-for-treatment-diagnostics